CLINICAL TRIAL: NCT04210830
Title: Comparison of Methods for Coagulation Analysis Between Rotem Sigma (Instrumentation Laboratory, Bedfort, MA, USA) and Quantra System (Hemosonics, Charlottesville, VA USA) in Cardiac Surgery
Brief Title: Comparison Two Point of Care Coagulation Monitoring Systems - the ROTEM Sigma and the Quantra Devic
Status: Completed | Type: Observational
Sponsor: Klinik Hirslanden, Zurich (Other)
Responsible Party: Principal Investigator, Werner Baulig, Prof. Dr. med., Klinik Hirslanden, Zurich
Other Study IDs: KlinikHirslande; NCT04310124 (obsolete NCT alias)
Record Dates: First submitted 2019-10-03; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Non Inferiority of the Quantra Device

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for Measurement the coagulation state of whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Quantra-Device — Point of Care Coagulation Monitoring System

SUMMARY:
Human Research Project Risk Category A. In this study no additional intervention or treatment are performed. The whole blood samples are taken from a routinely placed arterial catheter. The blood loss caused by the two additional blood samples is estimated with 2x 2.7ml. The Risk for the patients to participate in this study is minimal.

Clinical observational study of a point of care in vitro diagnostic device, the Quantra®system (Quantra), that received the CE Mark in April 2017 and is approved by the Swiss Medic for clinical use. The Quantra estimates the coagulation strength of whole blood by sonorheometry technology applying a series of ultrasound pulses to a whole blood sample and measuring its stiffness by returning echoes.

DETAILED DESCRIPTION:
The purpose of this study is to investigate to what extent the results of the Quantra corresponds to those of the ROTEM® Sigma (ROTEM). Additionally, the time required for delivery of final results (turnaround time) of all parameters of the Quantra will be examined. Significant differences in the turnaround time between both devices are of high interest as timing is a crucial factor in the diagnosis-based treatment.

Comparison of the coagulation process measurements in turnaround time and results of the ROTEM INTEM CT, HEPTEM CT, EXTEM A10 FIBTEM A10 with corresponding Quantra parameters such as CT, CTH, CTR, CS, PCS, FCS.

The primary aim of the study is to examine whether the two methods of hemostasis analysis are equivalent and how far they correlate.

Secondary aims are to examine the turnaround time of test results in both devices and to examine whether these results would have led to the same therapeutic decisions in a retrospective review of data.

For both devices following data is documented:

* Time for cartridge insertion
* Time first results available
* Time measurement finished

Parameters measured ROTEM Quantra

* INTEM CT Clot Time (CT)
* HEPTEM CT Heparinase Clot time
* (CTH)
* INTEM CT/HEPTEM CT Clot Time Ratio (CTR)
* EXTEM A10 Clot Stiffness (CS)
* FIBTEM A10 Fibrinogen Contribution
* to Clot Stiffness (FCS)
* EXTEM A10 - FIBTEM A10 Platelet Contribution to
* Clot Stiffness (PCS)

Blood loss estimated (mL/6h; mL/12h; mL/24 h) RCP transfused FFP packages transfused Platelet packages transfused Fibrinogen applied F XIII applied

Quantra clot stiffness values are expressed in hectoPascals (hPa), whereas corresponding ROTEM values are expressed as an amplitude in mm. The relationship between amplitude (A in mm) and shear modulus (G in Pascals) is not linear. For a proper comparison the ROTEM amplitude (mm) needs to be converted to Pascals by following formula:

G (Pascals) = (500 x A) / (100 - A),

as described by Solomon C et al, Anaesth Analg 2015; 121:868-78.

The Quantra data that are collected during the study are only observational and will not be used to guide therapeutic interventions

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cardiac surgery needing a cardiopulmonary bypass
* Age older than18 years
* Written consent of the participation after clarification about the study

Exclusion Criteria:

* No consent to participate
* No German comprehension
* Known coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Equivalence of the results of both devices | 1 Year
  Comparision of the results of the INTEM CT (R) with the Clot Time (Q)
Equivalence of the results of both devices | 1 Year
  HEPTEM CT (R) was compared with the Heparinase Clot ime (Q)
Equivalence of results of both devices | 1 Year
  INTEM CT/HEPTEM CT (R) was compared with the Clot Time Ratio (Q)
Equivalence of results of both devices | 1 Year
  EXTEM A10 (R) was compared with the Clot Stiffness (Q)
Equivalence of results of both devices | 1 Year
  FIBTEM A10 (R) was compared with the Fibrinogen Contribution to Clot Stiffness (Q)
Equivalence of results of both devices | 1 Year
  Difference of EXTEM A10 and FIBTEM A10 (R) was compared with the Platelet Contribution to Clot Stiffness (Q)

SECONDARY OUTCOMES:
Turnaround time of the measurements | 1 Year
  Time from taking the blood sample until introduction the Cartridge, in seconds
Turnaround time of the measurements | 1 Year
  Time from Insertion the Cartridge until the first plotted result
Turnaround time of the measurements | 1 Year
  Time from insertion the Cartridge until the all results are plotted

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik Im Park, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baulig W, Akbas S, Schutt PK, Keul W, Jovic M, Berdat P, von Felten S, Steigmiller K, Ganter MT, Theusinger OM. Comparison of the resonance sonorheometry based Quantra(R) system with rotational thromboelastometry ROTEM(R) sigma in cardiac surgery - a prospective observational study. BMC Anesthesiol. 2021 Oct 28;21(1):260. doi: 10.1186/s12871-021-01469-5. PMID 34711167